CLINICAL TRIAL: NCT01393756
Title: A Phase Ib/II Study of Escalating Doses of Revlimid in Association With R-CHOP (R2-CHOP) in the Treatment of B-cell Lymphoma
Brief Title: Revlimid Dose 25 mg in Association With (R-CHOP) in the Treatment Follicular Lymphoma
Acronym: R2-CHOP2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2-CHOP2
Record Dates: First submitted 2011-07-04; First posted 2011-07-13 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide dose 25 mg (Experimental)
  Interventions: Drug: Lenalidomide and R-CHOP

INTERVENTIONS:
Drug: Lenalidomide and R-CHOP — Lenalidomide dose administered orally during 14 days in combination with 6 courses of fixed doses of R-CHOP 21.
  Other Names: R2-CHOP2

SUMMARY:
The purpose of the study is to assess the efficacy of the association of Lenalidomide (Revlimid) and R-CHOP (Rituximab, Cyclophosphamide, Doxorubicin, vincristine and Prednisone) in a population of patients with follicular lymphoma as measured by the response rate at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with follicular lymphoma, (WHO) grade 1, 2 or 3a with at least one of the following signs requiring initiation of treatment:

  * Bulky disease according to the GELF criteria: nodal or extra-nodal mass >7cm in its greater diameter
  * B symptoms
  * Elevated serum (LDH) or beta 2-microglobulin
  * Involvement of at least 3 nodal sites (each >3cm)
  * Symptomatic spleen enlargement
  * Compressive syndrome
  * Pleural or peritoneal effusion
* Aged from 18 to 70 years
* WHO performance status 0, 1 or 2
* Signed inform consent
* Life expectancy of ≥ 90 days (3 months).
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL not more than 3 days from the start of study drug and must either commit to continued abstinence from heterosexual intercourse (and confirmed on a monthly basis) or begin one effective method of birth control, at least four weeks before she starts taking lenalidomide, and maintain that method throughout the entire duration of study drug therapy (including dose interruptions), and for four weeks after the end of study treatment with lenalidomide, even if she has amenorrhea. FCBP must also agree to pregnancy testing at least every three weeks and must be counseled at a minimum of every three weeks about pregnancy precautions and risks of fetal exposure.
* Men must agree not to father a child and agree to use a condom throughout study drug therapy, during any dose interruption, and for one week after cessation of study drug therapy, if their partner is pregnant or of child bearing potential. Men must also agree not to donate semen during study drug therapy and for one week after end of study drug therapy. Men must be counseled at a minimum of every 4 weeks about pregnancy precautions and risks of fetal exposure.
* All subjects must abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
* Agree not to share study drug with another person and to return all unused study drug to the investigator.

  * A female patient is considered to have childbearing potential unless she meets at least one of the following criteria 1) Age ≥ 50 years and naturally amenorrhoeic for ≥ 1 year (amenorrhoea following cancer therapy does not rule out childbearing potential); or 2) Premature ovarian failure confirmed by a specialist gynaecologist or 3) Previous bilateral salpingo-oophorectomy (BSO), or hysterectomy, or 4) XY genotype, turner syndrome, uterine agenesis.

Exclusion Criteria:

* Previous treatment with immunotherapy or chemotherapy:

  * Chlorambucil or Cyclophosphamide per os alone during less than 6 months, if stopped more than one year before inclusion
  * Rituximab alone during less than three months, if stopped more than one year before inclusion
* Previous radiotherapy except if localized to one lymph node area
* Other type of lymphomas: Burkitt, T cell, lymphocytic, CD 20 negative
* Central nervous system or meningeal involvement
* Contraindication to any drug contained in the chemotherapy regimen
* (HIV) disease, active hepatitis B or C
* Any serious active disease or co-morbid medical condition (according to investigator's decision)
* Any of the following laboratory abnormalities.

  * Absolute neutrophil count (ANC) < 1,500 cells/mm3 (1.5 x 109/L).
  * Platelet count < 100,000/mm3 (100 x 109/L).
  * Serum (SGOT/AST) or (SGPT/ALT) 5.0 x upper limit of normal (ULN).
  * Serum total bilirubin > 2.0 mg/dL (34 µmol/L), except in case of hemolytic anemia.
* Calculated creatinine clearance (Cockcroft-Gault formula) of < 50 mL /min
* Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 3 years
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females.
* Prior ≥ Grade 3 allergic reaction/hypersensitivity to thalidomide.
* Prior ≥ Grade 3 rash or any desquamating (blistering) rash while taking thalidomide.
* Subjects with ≥ Grade 2 neuropathy.
* Prior use of lenalidomide.
* Use of any standard or experimental anti-cancer drug therapy within 28 days of the initiation (Day 1) of study drug therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-12; Primary Completion 2013-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Complete Response Rate (CR+CRu) | at the end of complete treatment, average of 24 weeks

SECONDARY OUTCOMES:
Overall survival | from the date of inclusion, average of 6 years
Duration of response | from the date of first documentation of a response, average of 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hervé TILLY, Professeur, Principal Investigator — Lymphoma Study Association
Locations (24):
- France (24):
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CHU de DIJON, Dijon
  - Chru Lille, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital Notre Dame de Bon Secours, Metz
  - Hôpital Saint Eloi, Montpellier
  - CHU de NANTES, Nantes
  - Hôpital Saint Antoine, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - Hôpital Necker, Paris
  - Institut Curie, Paris
  - Hôpital St Louis, Paris
  - Chu Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Hôpital Robert Debré, Reims
  - Hôpital Pontchaillou, Rennes
  - Centre Henri BECQUEREL, Rouen
  - Hôpital René Huguenin, Saint-Cloud
  - Chu Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tilly H, Morschhauser F, Casasnovas O, Molina TJ, Feugier P, Gouill SL, Haioun C, Tournilhac O, Bouabdallah R, Gabarre J, Lamy T, Cabecadas J, Becker S, Jardin F, Mounier N, Salles G; Lymphoma Study Association. Lenalidomide in combination with R-CHOP (R2-CHOP) as first-line treatment of patients with high tumour burden follicular lymphoma: a single-arm, open-label, phase 2 study. Lancet Haematol. 2018 Sep;5(9):e403-e410. doi: 10.1016/S2352-3026(18)30131-5. PMID 30172345
- See also: Lymphoma Study Association LYSA — http://www.lysa-lymphoma.org/